CLINICAL TRIAL: NCT01030302
Title: An Observational, Prospective Analysis of Retreatment With Bortezomib for Multiple Myeloma
Brief Title: A Retreatment Study With Bortezomib for Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015814; 26866138MMY4039 (Other: Janssen Korea, Ltd.); BORKOR5021 (Other: Janssen Korea, Ltd.)
Record Dates: First submitted 2009-10-29; First posted 2009-12-11 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Multiple Myeloma
Keywords: Bortezomib retreatment; Velcade; Proteasome inhibitor; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 001: bortezomib injection into a vein 1.3 mg/m2 twice a week for 21 days
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — bortezomib injection into a vein 1.3 mg/m2 twice a week for 21 days

SUMMARY:
The purpose of this study is to monitor such factors as a past history, a previous history of drug use, the degree of response to initial treatment, the frequency of previous therapies, age, Eastern Cooperative Oncology Group (ECOG) performance status, which is used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis, before the bortezomib re-treatment, the concomitant drugs that are used for re-treatment and the pattern of treatment in patients with multiple myeloma who were re-treated with injectable bortezomib.

DETAILED DESCRIPTION:
It will be essential to obtain the Korean clinical data about the efficacy and safety of the re-treatment with bortezomib as well as to analyze its actual pattern. The current trial is a prospective, multi-center, Phase 4, observational study that will be conducted to collect such demographic data as a past history, a previous history of drug use, the degree of responses to initial treatment, the frequency of previous therapies, age, Eastern Cooperative Oncology Group (ECOG) performance status, the concomitant drugs that are used for re-treatment and the pattern of treatment for patients with multiple myeloma and who were re-treated with injectable bortezomib. Also safety data will be collected. Observational Study -No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma
* Patients who were treated with bortezomib monotherapy or bortezomib combination therapy
* Patients who relapsed after >= six months interval since last dose of bortezomib
* Patients who had a treatment response of higher than partial remission (PR) to the previous bortezomib therapy
* Patients who were fully aware of the objectives and essential procedures of the current trial and then submitted a written informed consent declaring that they will voluntarily participate in the current trial

Exclusion Criteria:

* The current presence of or a past history of hypersensitivity to bortezomib or its constituents
* Severe hepatic dysfunction (AST or ALT at first use>= x 5 upper normal)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients who are scheduled to be re-treated with bortezomib for the recurrence of multiple myeloma and who have submitted a written informed consent to provide their personal data in relation to their former, prescribed use of bortezomib for the treatment of multiple myeloma in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To monitor such factors as a past history, a previous history of drug use, the degree of responses to initial treatment, the frequency of previous therapies, age, the concomitant drugs that are used for re-treatment and the pattern of treatment. | 6-12 months

SECONDARY OUTCOMES:
Adverse events | at the end of every 3 week cycle
Overall response rate | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

REFERENCES:
- See also: An Observational, Prospective Analysis of Retreatment with Bortezomib for Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=333&filename=CR015814_CSR.pdf